CLINICAL TRIAL: NCT02104349
Title: Mindfulness Meditation for Spine Surgery Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Arthur L Jenkins, Associate Clinical Professor, Neurosurgery, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 12-1322
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Meditation; Spine Surgery; Pain, Postoperative
Keywords: spine surgery; post op pain management
MeSH Terms: conditions — Pain, Postoperative | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness meditation (Experimental): Subjects who are instructed on use of the mindfulness meditation technique
  Interventions: Behavioral: Mindfulness meditation
- Control (No Intervention): Subjects will receive standard surgery treatment without any mindfulness intervention.

INTERVENTIONS:
Behavioral: Mindfulness meditation — One hour training with mindfulness instructor. Listening to mindfulness CD twice a day for 2 weeks prior to spine surgery. Post-operative practice will be at least 1 track per day.
  Arms: Mindfulness meditation

SUMMARY:
The objective of this study is to evaluate the effect of mindfulness meditation technique on post-operative pain of spine surgery subjects. Subjects will participate in a 6-week mindfulness meditation program, beginning two weeks prior to spine surgery. The investigators are interested in determining if this intervention improves the ability to tolerate pain and reduces anxiety, thus reducing the need for prescribed analgesics and narcotics. The meditation intervention will be compared against a control group consisting of subjects that will undergo music therapy during the same period of time.

DETAILED DESCRIPTION:
Mind body therapies which induce relaxation through the use of imagery and meditation, are being increasingly sought as treatments to assist individuals cope with stress and chronic illness. These holistic therapies have become accepted by both physicians and patients because of the recent emerging body of evidence supporting their effectiveness for a variety of physical and psychological conditions. In the case of holistic (or integrative) practices used to alleviate pain, the infrequency of adverse effects makes them particularly attractive to physicians who have become wary of the risks of prescription narcotics.

Pain medications, though they provide immediate relief, have many noted adverse side effects. These include respiratory depression, decreased heart rate and in extreme cases of misuse, death. These medications are especially prone to abuse by patients, even after their initial pain subsides. Overdosing from prescription pain killers has become a significant cause of accidental death, and providers are seeking alternative treatments for pain for their patients that do not carry this risk.

A significant body of research has investigated the benefits of meditation for a wide variety of physical and psychological conditions . However, clinical evidence for the efficacy of meditation for reducing pain is sparse, although some research suggests the mechanisms of this possible benefit , Mindfulness-Based Stress Reduction (MBSR) is a mindfulness intervention which is currently used in over 500 clinical sites around the world for patients with a wide variety of clinical problems, including pain. MBSR was developed by Jon Kabat Zinn at the University of Massachusetts in the 1970s. It is derived from the Oriental traditions of Zen Buddhism, yet free from its religious roots. It is supported by over 30 years of research that substantiate its positive effects on numerous ailments, including stress , chronic pain , anxiety and depression .

The key concept in mindfulness meditation involves learning how to observe the thoughts that enter one's mind without the passing of judgment and by keeping the focus on breathing or another constant. This is called "detached observation". The mechanisms at work are unknown but are thought to be the meditation facilitating the tuning out of distractions by learning to maintain and control attention.

The process of mindfulness meditation entails sitting in a quiet location and comfortable position with one's eyes closed. Individuals are instructed to relax and focus on their breathing, or another chosen object of attention, such as parts of the body in the body scan, body movements in mindful movement, or the act of walking in walking meditation. While the mind may wander and numerous thoughts, worries or concerns may arise, the individual learns to non-self-critically acknowledge the shift in attention, and return to the chosen object of attention. Over time, increased attentional control and awareness of mental events leads to the ability to respond more positively and less reactively to stressful events, including pain.

An early study of MBSR for chronic pain patients found that, after a 10-week training program, participants demonstrated statistically significant reductions in pain, negative body image, pain-related reductions in activity, anxiety, and depression, compared with a control group5.

Whereas the benefit of MBSR for pain has been suggested by existent research, the fact that it is an 8-week course requiring participation on a weekly basis in 2 ½ hour classes, with daily practice at home of 30-45 minutes, may limit its accessibility to some patients. This study seeks to identify an intervention that may be widely used by participants with both acute and chronic pain.

Open Focus technique is a specific mindfulness-based practice developed by Les Fehmi, PhD, of Princeton, NJ. It guides practitioners to modify their attention in ways that have been shown to promote relaxation and pain reduction, as measured by brain wave activity .

Additionally, recent research has reported actual physical and structural changes in the brain with long term practice of meditation. Benefits of mindfulness meditation appear to have a neuroplastic effect on the brain. Studies among those practicing meditation have demonstrated a change in the mass of grey matter as well as an increase in brain connectivity . The structural changes in the brain include an increased density of grey matter in the hippocampus, which is a region involved in the process of learning and memory. In addition, a decrease in density in the amygdala was noted; this region plays a role in stress and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Patients that will undergo spine surgery including: single level lumbar fusion, posterior cervical laminectomy fusion, cervical laminaplasty

Exclusion Criteria:

* Patients with scheduling conflicts that will render them unable to follow the weekly mindfulness mediation instruction.
* Patients with depression (established during the screening questionnaire)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 2 weeks prior to surgery
  Visual Analog Scale (VAS) to measure pain: a measure of "no pain" to "Worst pain imaginable" along a line. Participants will be asked to mark the level of their pain along the line. Total score ranges 0-10, with higher scores indicating higher levels of pain.
Change in Visual Analog Scale (VAS) | Baseline up to 6 weeks
  Visual Analog Scale (VAS) to measure pain: a measure of "no pain" to "Worst pain imaginable" along a line. Participants will be asked to mark the level of their pain along the line.

SECONDARY OUTCOMES:
Oswestry Disability Index | 2 weeks prior to surgery
  It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5. If a patient marks more than one statement in a question, the highest scoring statement is recorded as a true indication of disability.
Oswestry Disability Index | baseline up to 6 weeks
  It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5. If a patient marks more than one statement in a question, the highest scoring statement is recorded as a true indication of disability.
Perceived Stress Scale | 2 weeks prior to surgery
  A 10-item self-report scale that was developed to measure the degree to which situations in one's life are appraised as stressful. Total score ranges 0-40, with higher scores indicating higher levels of perceived stress.
Perceived Stress Scale | baseline up to 6 weeks
  A 10-item self-report scale that was developed to measure the degree to which situations in one's life are appraised as stressful. Total score ranges 0-40, with higher scores indicating higher levels of perceived stress.
Hospital Anxiety and Depression Scale | 2 weeks prior to surgery
  14-items scale with responses scored from 0-3, scores for each subscale from 0 (normal) to 21 (severe symptoms). Scores for the entire scale is 0 to 42, with higher score indicating more distress.
Hospital Anxiety and Depression Scale | baseline up to 6 weeks
  14-items scale with responses scored from 0-3, scores for each subscale from 0 (normal) to 21 (severe symptoms). Scores for the entire scale is 0 to 42, with higher score indicating more distress.
Muscle Relaxer Dosage | 2 weeks prior to surgery
  Pre-Operative Muscle Relaxer dosage
Antidepressant Dosage | 2 weeks prior to surgery
  Pre-Operative Antidepressant dosage
Neuropathics Dosage | 2 weeks prior to surgery
  Pre-Operative Neuropathics dosage
Narcotics Dosage | 2 weeks prior to surgery
  Pre-Operative Narcotics dosage
NSAIDS Dosage | 2 weeks prior to surgery
  Pre-Operative NSAIDS dosage
Muscle Relaxers dosage | baseline up to 6 weeks
  Post-Operative Muscle Relaxers dosage
Neuropathics dosage | baseline up to 6 weeks
  Post-Operative Neuropathics dosage
Narcotics dosage | baseline up to 6 weeks
  Post-Operative Narcotics dosage
NSAIDS dosage | baseline up to 6 weeks
  Post-Operative NSAIDS dosage

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Jenkins, III, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States